CLINICAL TRIAL: NCT00408161
Title: Contingency Management for Chronic Recidivist Alcohol-Dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-PET03510; NIH Grant P50-AA03510
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Dependence
Keywords: Contingency Management; Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): prize contingency management (CM) plus standard case management treatment -- patients earn the chance to win prizes by submitting negative breath samples and by complying with steps toward treatment goals
  Interventions: Behavioral: Contingency Management
- 2 (Active Comparator): standard case management treatment
  Interventions: Behavioral: standard case management treatment

INTERVENTIONS:
Behavioral: Contingency Management — prize contingency management (CM) -- 6-month treatment plus standard case management treatment and follow-ups at 9, 12, and 18 months after intake
  Other Names: CM
  Arms: 1
Behavioral: standard case management treatment — 6-month treatment standard case management treatment, and follow-ups scheduled at 9, 12, and 18 months after intake.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of prize contingency management (CM) in reducing in-patient detoxification services for chronic recidivist alcohol-dependent patients.

DETAILED DESCRIPTION:
This study evaluates the efficacy of prize contingency management (CM) in reducing in-patient detoxification services for chronic recidivist alcohol-dependent patients. 116 alcohol-dependent patients who have received 4 or more alcohol detoxifications in a calendar year will be randomly assigned to one of two 6-month treatment conditions: standard case management treatment, or standard case management treatment plus CM. In the CM condition, patients earn the chance to win prizes by submitting negative breath samples and by complying with steps toward treatment goals, such as attending outpatient substance abuse treatment services, attending appointments with low income housing programs, or complying with outpatient psychiatric treatment. Treatment services received, alcohol and drug use, psychosocial functioning, and HIV risk behaviors will be measured pre-treatment and at months 1, 3, and 6 (post-treatment), and at follow-ups scheduled for 9, 12, and 18 months after intake.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Four or more inpatient alcohol detoxifications in the previous 12 months
* current diagnosis of DSM-IV alcohol dependence

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
number of detoxifications | 9, 12, and 18 months after intake
objective alcohol use | 9, 12, and 18 months after intake
self-reported alcohol use | 9, 12, and 18 months after intake

SECONDARY OUTCOMES:
ASI composite scores | 9, 12, and 18 months after intake
BSI scores | 9, 12, and 18 months after intake
HRBS scores | 9, 12, and 18 months after intake
objective drug use | 9, 12, and 18 months after intake

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States